CLINICAL TRIAL: NCT03164473
Title: MAINtenance of Remission With RITuximab Versus Azathioprine for Patients With Newly-diagnosed or Relapsing Eosinophilic Granulomatosis With Polyangiitis. A Prospective, Randomized, Controlled, Double-blind Study: the MAINRITSEG Trial
Brief Title: Maintenance of Remission With Rituximab Versus Azathioprine for Newly-diagnosed or Relapsing Eosinophilic Granulomatosis With Polyangiitis.
Acronym: MAINRITSEG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French Vasculitis Study Group (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P150922; 2016-000627-53 (EudraCT Number)
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Eosinophilic Granulomatosis With Polyangiitis
Keywords: Eosinophilic granulomatosis with polyangiitis in remission; double-blind randomized controlled trial; maintenance therapy; rituximab versus azathioprine; vasculitis remission; asthma control; rhinosinusal manifestations control; glucocorticoid therapy reduction/withdrawal; steroid sparing effect; damage
MeSH Terms: conditions — Churg-Strauss Syndrome | interventions — Rituximab; Azathioprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab (Experimental): * pre-emptive 500-mg fixed-dose of IV rituximab every 6 months (total duration of 18 months = 4 infusions)
  * plus orally placebo-azathioprine for 24 months
  Interventions: Drug: Rituximab; Drug: Placebo-azathioprine
- Azathioprine (Active Comparator): * standard maintenance oral azathioprine therapy (2 mg/kg/day) for 24 months
  * plus 4 placebo-rituximab infusions given every 6 months for 18 months
  Interventions: Drug: Azathioprine; Drug: Placebo-rituximab

INTERVENTIONS:
Drug: Rituximab — pre-emptive 500-mg fixed-dose of IV rituximab every 6 months (total duration of 18 months = 4 infusions)
  Arms: Rituximab
Drug: Azathioprine — oral tablets : 2 mg/kg/day for 24 months
  Arms: Azathioprine
Drug: Placebo-rituximab — 4 infusions for 18 months
  Arms: Azathioprine
Drug: Placebo-azathioprine — oral tablets for 24 months
  Arms: Rituximab

SUMMARY:
The purpose of this study is to investigate, after achievement of remission, the efficacy of rituximab compared with azathioprine maintenance therapy on duration of remission, in patients with relapsing or newly-diagnosed Eosinophilic granulomatosis with polyangiitis EPGA receiving standard of care therapy including glucocorticoid therapy reduction/withdrawal.

DETAILED DESCRIPTION:
Rituximab, an anti-CD20 monoclonal antibody, has been shown to be as effective as cyclophosphamide to induce GPA and MPA remission, with an acceptable safety profile, leading to its registration by the FDA and EMA as remission-induction therapy in these patients.

In addition, the MAINRITSAN trial has demonstrated that 500 mg rituximab given every 6 months for 18 months was significantly more effective than azathioprine standard of care to maintain remission in patients with GPA or MPA, with a similar profile of tolerance.

EGPA patients were excluded from these trials. Long-term studies have shown that only 29% of EGPA patients achieved long-term remission and that relapses occurred in more than 40% of them, leading to high cumulative morbidity and damage. Moreover, most patients cannot be weaned off corticosteroids due to asthma and rhino-sinusal manifestations, even after vasculitis remission.

However, recent retrospective series indicated that rituximab may also be an effective remission induction and maintenance agent in refractory or relapsing EGPA. REOVAS, the first randomized controlled trial with rituximab as induction therapy in EGPA, has started within the French Vasculitis Study Group network.

The MAINRITSEG trial is a phase III, comparative, multicenter, randomized, double-blind, double-dummy and superiority trial, comparing pre-emptive low-dose rituximab-based regimen with azathioprine standard therapy, for the remission maintenance in newly-diagnosed or relapsing EGPA.

Patients, with newly diagnosed or relapsing EGPA, after achievement of remission, will be randomized in a 1:1 ratio to receive:

* Standard regimen: maintenance oral azathioprine (2 mg/kg/day) for 24 months. This control group will receive conventional therapy plus 4 infusions of placebo-rituximab (every 6 months for 18 months)
* Experimental regimen: pre-emptive 500-mg fixed-dose of rituximab every 6 months for 18 months (4 infusions). This group will receive intravenous rituximab plus orally placebo-azathioprine for 24 months.

All patients will receive standard of care therapy including glucocorticoid therapy reduction/withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of EGPA according to Lanham and/or ACR 1990 criteria and/or Revised Chapel Hill Nomenclature and/or MIRRA study inclusion criteria
* 18 years of age or more
* with newly-diagnosed EGPA or after a vasculitis flare and remission achieved within the past year
* independently of ANCA status
* within 30-360 days following achievement of vasculitis remission (corresponding to a Birmingham Vasculitis Activity Score (BVAS)=0) achieved with an induction regimen including the one used in the REOVAS trial: either CS alone or in association with CYC (total dose ranging from 4.5-10 g for patients <65 years old and from 3-10g for patients ≥65 years old) or RTX (2 x 1g (D1, D15) or 4 weekly 375 mg/m2).
* with a stable prednisone dose for 30 days or no more prednisone
* after oral immunosuppressive drug cessation if started at remission.
* Patients included in the REOVAS trial and achieving remission can be included at month 12 visit if they fulfil the other criteria
* Patients able to give written informed consent prior to participation in the study.
* Affiliation with a mode of social security (profit or being entitled).

Exclusion Criteria:

* patients with GPA, MPA or other vasculitides
* patients with vasculitis not in remission defined as a BVAS >0
* acute or chronic active infections (including HIV, HBV or HCV)
* active or recent cancer ( <5 years), except basocellular carcinoma and low activity prostatic cancer controlled by hormonal treatment
* severe heart failure (New York Heart Association Class IV) or severe, uncontrolled cardiac disease
* pregnant women and lactation
* patients with childbearing potential will have reliable contraception for all the duration of the study and another 12 months after. Women are considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient
* men who refuse to use effective method of contraception (condom) from the date of consent through the end of the study
* patients who had already been treated with rituximab before the last relapse/flare
* patients who have been treated with rituximab with a different induction regimen than 2 x 1g (D1, D14) or 4 weekly 375 mg/m2 infusions
* hypersensitivity to a monoclonal antibody or biologics
* contraindication to rituximab or azathioprine
* other uncontrolled diseases, including drug or alcohol abuse, severe psychiatric diseases, that could interfere with participation
* patients included in other investigational therapeutic study within the previous 3 months except in the REOVAS trial, after which patients achieving remission can be included if they fulfil the other criteria
* patients suspected not to be observant to the proposed treatments
* white blood cell count ≤4,000/mm3
* platelet count ≤100,000/mm3
* ALT or AST level >3 times the upper limit of normal
* patients not able to stop allopurinol and febuxostat which may enhance azathioprine toxicity
* patients unable to give written informed consent prior to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Duration of remission in weeks | 28 months
  accrued number of weeks where a patient remains in remission with BVAS=0 and prednisone dose ≤7.5 mg/day

SECONDARY OUTCOMES:
proportion of patients remaining in remission with a BVAS=0 and prednisone dose ≤7.5 mg/day | 28 months
Accrued number of weeks where a patient remains in remission with BVAS=0 and prednisone dose ≤4 mg/day | 28 months
proportion of patients remaining in remission with a BVAS=0 over the 28 months study period | 28 months
proportion of participants who achieved remission of vasculitis (BVAS = 0) while receiving prednisone at a dose of 4.0 mg or less per day at month 6 | 6 months
proportion of participants who achieved remission of vasculitis (BVAS = 0) while receiving prednisone at a dose of 4.0 mg or less per day at month 12 | 12 months
proportion of participants who achieved remission of vasculitis (BVAS = 0) while receiving prednisone at a dose of 4.0 mg or less per day at month 18 | 18 months
proportion of participants who achieved remission of vasculitis (BVAS = 0) while receiving prednisone at a dose of 4.0 mg or less per day at month 28 | 28 months
proportion of patients with at least one vasculitis relapse (major, minor, either) | 28 months
proportion of patients with at least one clinically significant asthma/rhino-sinusal exacerbation | 28 months
  defined as a worsening of asthma/rhino-sinusal disease leading to the doubling (or more) of the existing maintenance dose of corticosteroids for 3 or more days or hospital admission or an emergency department visit.
time to first vasculitis relapse | 28 months
time to first clinically significant asthma/rhino-sinusal exacerbation | 28 months
  defined as a worsening of asthma/rhino-sinusal disease leading to the doubling (or more) of the existing maintenance dose of corticosteroids for 3 or more days or hospital admission or an emergency department visit.
variation of the obstructive pulmonary disease | 28 months
  assessed by change of FEV1 at pulmonary function tests after use of a bronchodilator
prednisone dose at months 6, 12, 18, 24 and 28, and area under the curve over the 28 month study period | 28 months
proportion of patients with adverse events | 28 months
proportion of patients with serious adverse events | 28 months
proportion of patients with selected severe adverse events including grade 3 or 4 adverse effects (Common Terminology Criteria for Adverse Events) | 28 months
  necessitating hospitalization, all cause deaths, cancers or infusion reactions (within 24 hours of infusion) that contraindicated further infusions
number and causes of deaths over the 28 month study period | 28 months
damage assessed by the mean variation of the Vasculitis Damage Index (VDI) | 28 months
quality of life assessed by the mean variation of the SF-36 | 28 months
disability assessed by the mean variation of the Health Assessment Questionnaire (HAQ) | 28 months
number of days of hospitalization | 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Terrier, Study Chair — National Referral Center for Rare Systemic Autoimmune Diseases - Hôpital Cochin
Locations (1):
- Hôpital Cochin, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No